CLINICAL TRIAL: NCT04145219
Title: A One-year Placebo-controlled Phase III Trial Evaluating the Efficacy and Safety of the House Dust Mite (HDM) SLIT-tablet in Children (5-11 Years of Age) With HDM Allergic Rhinitis/Rhinoconjunctivitis With or Without Asthma
Brief Title: House Dust Mite Allergy Trial In Children
Acronym: MATIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-12
Record Dates: First submitted 2019-10-11; First posted 2019-10-30 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Allergic Rhinitis Due to Dermatophagoides Farinae; Allergic Rhinitis Due to Dermatophagoides Pteronyssinus; Allergic Rhinitis Due to House Dust Mite
Keywords: Allergic rhinitis; HDM; pediatric
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): HDM SLIT-tablet plus allergy and asthma rescue medication
  Interventions: Biological: Sublingual allergy immunotherapy tablet
- Placebo (Placebo Comparator): Placebo oral tablet plus allergy and asthma rescue medication
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Sublingual allergy immunotherapy tablet — For daily administration (1 tablet per day)
  Other Names: Acarizax; Odactra
  Arms: Active treatment
Other: Placebo — For daily administration (1 tablet per day)
  Other Names: Placebo sublingual tablet
  Arms: Placebo

SUMMARY:
A research study of how house dust mite tablets work compared to placebo in children aged between 5 and 11 years and who have allergy to house dust mites (MATIC)

DETAILED DESCRIPTION:
The trial aims to demonstrate efficacy of the House Dust Mite SLIT-tablet compared to placebo in children (5-11 years of age) with House Dust Mite allergic rhinitis based on the total combined rhinitis symptoms and medication score during the last 8 weeks of treatment.

In addition, the trial will evaluate safety and tolerability of the treatment, and assess whether treatment has an impact on asthma symptoms and medication use, immunological parameters, and rhinoconjunctivitis quality of life (QoL).

The trial is a randomised, parallel-group, double-blind, placebo-controlled multi-national phase III trial conducted in Europe and North America. The treatment period will be approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 5-11 years
* A clinical history of HDM AR/C (Allergic rhinitis/rhinoconjunctivitis) (with or without asthma) and with allergic rhinitis symptoms despite having received allergy pharmacotherapy during the previous year prior to screening
* Have a certain level of AR (Allergic rhinitis) symptoms on at least 8 of the last 14 days of the baseline period
* Use symptomatic medication for treatment of HDM allergic rhinitis during at least 8 of the last 14 days of the baseline period
* Positive skin prick test (SPT) and IgE (Immunoglobulin E) to D. pteronyssinus or D. farinae at screening
* Lung function ≥ 70% of predicted value

Exclusion Criteria:

* Sensitised and regularly exposed to perennial allergens
* Any nasal or pharyngeal condition that could interfere with the safety or efficacy evaluation
* Asthma requiring treatment with high dose of inhaled corticosteroid
* A relevant history of systemic allergic reaction

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1460 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antje Schuster, MD, Principal Investigator — Professor of Pediatrics, Düsseldorf University Hospital
Locations (112):
- United States (29):
  - Allergy & Asthma Specialists Medical Group and Research Center, Huntington Beach, California
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - Allergy & Asthma Medical Group and Research Center, A P.C., San Diego, California
  - Miami Clinical Research, Miami, Florida
  - Pensacola Research Consultants, Inc. d.b.a. Avanza Medical Research Center, Pensacola, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - GCP, Global Clinical Professionals, St. Petersburg, Florida
  - Aeroallergy Research Labs of Savannah, Inc., Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Deaconess Clinic Allergy, Evansville, Indiana
  - PMG Research of McFarland Clinic, Ames, Iowa
  - Clinical Research Institute, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Clinical Research of The Ozarks Inc, Warrensburg, Missouri
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Allergy & Asthma Associates of Monmouth City, Little Silver, New Jersey
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - The Children's Research Institute, Department of Pediatrics, University of North Carolina Children's Hospital, Chapel Hill, North Carolina
  - UNC Children's Raleigh, Raleigh, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Oklahoma Institute of Allergy & Asthma Clinical Research, LLC, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - The Corvallis Clinic, Corvallis, Oregon
  - West Ashley office: Charleston Allergy & Asthma, Charleston, South Carolina
  - ADAC Research, PA, Greenville, South Carolina
  - Charleston Allergy & Asthma, Summerville, South Carolina
  - Biogenics Research Institute, San Antonio, Texas
  - Allergy, Asthma & Sinus Center, S.C., Greenfield, Wisconsin
- Bulgaria (11):
  - Multiprofile Hospital for active treatment, Department of Pediatrics, Gabrovo
  - Multiprofile Hospital for Active Treatment, Department of Pediatrics, Kyustendil
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD, Plovdiv
  - Multiprofile Hospital for Active Treatment, Department of pneumology and phthisiatrics, Razgrad
  - Outpatient Clinic for individual practice for specialized outpatient medical care in Allergology, Razgrad
  - Specialized Hospital For Active Treatment of Pneumo - Phtisiatric Diseases Dr Dimitar Gramatikov - Ruse, Rousse
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda, EAD, Clinic in Pediatrics, Sofia
  - Sv. Vratch and Sv.Sv. Kuzma i Damian, Sofia
  - Alitea-Med-Medical-Center, Sofia
  - Diagnostic-Consultative center Ritam TR, Stara Zagora
- Canada (10):
  - Halton Pediatric Allergy, Burlington
  - Triple A Lab, Hamilton
  - Kingston General Hospital - Division of Allergy & Immunology, Kingston
  - CHU Ste-Justine, Montreal
  - The Montreal Children's Hospital, Montreal
  - Niagara Clinical Research, Niagara Falls
  - Gordon Sussman Clinical Research, Inc., North York
  - Clinique spécialisée en allergie de la capitale, Québec
  - Hospital for Sick Children, Toronto
  - Joel Liem Medicine Professional Corporation, Windsor
- France (2):
  - Hôpital Morvan - Service de Pédiatrie, Brest
  - CHU de Montpellier - Service Pneumologie et Addictologie, Montpellier
- Germany (4):
  - Kinderarztpraxis Bramsche, Bramsche
  - HNO praxis - Dr Yury Yarin, Dresden
  - Klinikum der Johann-Wolfgang-Goethe Universität - Zentrum f. Kinder- u. Jugendmedizin, Frankfurt
  - GMAP/HNO am Neckar, Heidelberg
- Lithuania (5):
  - CD8 klinika, Kaunas
  - Siauliai Republican Hospital, Šiauliai
  - JSC Seimos gydytojas, Vilnius
  - Center of Allergy Diagnosis and Treatment, Vilnius
  - Inlita JSC, Santara KTC, Vilnius
- Poland (11):
  - Indywidualna Specjalistyczna Praktyka Lekarska Elzbieta Matusz, Gryfice
  - Specjalistyczna Praktyka Lekarska Dr n. med. Joanna Orlicz-Widawska, Katowice
  - Centrum Medyczne ALL-MED, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Poradnia Alergologiczna, Lodz
  - Alergotest s.c. Specjalistyczne Centrum Medyczne Andrzej Emeryk, Lublin
  - Centrum Alergologii Teresa Hofman Sp. z o.o., Poznan
  - Podkarpacki Ośrodek Pulmonologii i Alergologii Sp. z o.o., Rzeszów
  - Prywatny Gabinet Lekarski Malgorzata Pawlukiewicz, Rzeszów
  - IRMED Irena Wojciechowska, Warsaw
  - All-Med" Specjalistyczna Opieka Medyczna, Medyczny Instytut Badawczy Marek Jutel, Wroclaw
- Russia (16):
  - City Children's Hospital, Kolpino
  - Prof. V.F. Voino-Yasenetsky Krasnoyarsk State Medical University, Krasnoyarsk
  - NRC Institute of Immunology, Moscow
  - Moscow City Children's Hospital No 9, Moscow
  - City Сhildren's Сlinical Polyclinic No5, Perm
  - I.P. Pavlov Ryazan State Medical University, Ryazan
  - Medical Technologies" Ltd., Saint Petersburg
  - City Children's Polyclinic No44, Saint Petersburg
  - ArsVitae Severo-Zapad LLC, Saint Petersburg
  - North-Western State Medical University named after I.I. Mechnikov, Ministry of Public Health of Russian Federation, Saint Petersburg
  - Сurator LLC, Saint Petersburg
  - City Children's Polyclinic No45, Saint Petersburg
  - Сity Children's Polyclinic No 35, Saint Petersburg
  - Smolensk State Medical University, Smolensk
  - Scientific Medical Center for General Therapy and Pharmacology, Stavropol
  - Regional Children's Hospital, Tomsk
- Slovakia (4):
  - Alersa, s.r.o, Ambulancia klinickej alergológie a imunológie, Košice
  - Ambulancia klinickej imunologie a alergologie, Levice
  - ALFA EL, Imunoalergologická ambulancia, Poprad
  - Ambulancia klinickej imunologie a alergologie, Šurany
- Spain (6):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera
  - Hospital de Sagunto, Sagunto
  - Hospital de Sagunto, Valencia
  - Hospital la Plana, Villarreal
- Ukraine (14):
  - Chernivtsi Regional Children's Clinical Hospital, Department of Pediatrics and Children's Infectious Diseases, Chernivtsi
  - Clinical Emergency Hospital" of Dnipro City Council, Department of Pediatric Allergology at the Allergology Center, Dnipro
  - Dnipro City Children's Municipal Clinical Hospital #2, Dnipro
  - City Children's Clinic № 16" of Kharkiv City Council, Kharkiv
  - City Children's Clinical Hospital # 19" of Kharkiv City Council, Kharkiv
  - Kryvyi Rih City Clinical Hospital #8'' of Kryvyi Rih City Council, Department of Pediatric Pulmonology; State Institution "Dnipropetrovsk Medical Academy of the Ministry of Health of Ukraine, Kryvyi Rih
  - O.S. Kolomiychenko Institute, Center of Allergic Diseases of Upper Respiratory Ways and Ear, Kyiv
  - State Institution Phthisiology and Pulmonology Institute named after F.G. Yanovskyy of NAMS of Ukraine, Kyiv
  - Institute of Pediatrics, Obstetrics and Gynecology named after Academician O. M. Lukianova of the National Academy of Medical Sciences of Ukraine, Kyiv
  - Communal Nonprofit Enterprise "Lviv City Children's Clinical Hospital", Allergology Department, Lviv City Children's Allergology Center, Lviv
  - Children's Clinical Hospital of Poltava Regional Council, Poltava
  - Regional Children Clinical Hospital, Infectious-Diagnostic Department, Sumy
  - Regional Children's Clinical Hospital of Vinnytsia Regional Council, Vinnytsia
  - City Children's Hospital #5" of Zaporizhzhya City Council, Allergology Department, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuster A, Caimmi D, Nolte H, Novakova S, Mikler J, Foss-Skiftesvik MH, Osterdal AS, Emeryk A, Gagnon R, Pfaar O. Efficacy and safety of SQ house dust mite sublingual immunotherapy-tablet (12 SQ-HDM) in children with allergic rhinitis/rhinoconjunctivitis with or without asthma (MT-12): a randomised, double-blind, placebo-controlled, phase III trial. Lancet Reg Health Eur. 2024 Nov 26;48:101136. doi: 10.1016/j.lanepe.2024.101136. eCollection 2025 Jan. PMID 39678704
- [Derived] Field K, Blaiss MS. Sublingual Versus Subcutaneous Immunotherapy for Allergic Rhinitis: What Are the Important Therapeutic and Real-World Considerations? Curr Allergy Asthma Rep. 2020 Jun 16;20(9):45. doi: 10.1007/s11882-020-00934-4. PMID 32548677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial randomized 1460 participants from 95 sites in 11 countries (Bulgaria, Canada, France, Germany, Lithuania, Poland, Russia, Slovakia, Spain, Ukraine, United States).
Pre-assignment Details: The trial randomized 1460 participants. Two participants in the 12 SQ-HDM group were randomized in error and did not receive study treatment, hence the number of participants that started (who were randomized and treated) is 1458.
Groups:
- HDM SLIT-tablet (12 SQ-HDM): Rhinitis/rhinoconjunctivitis rescue medication as needed, plus daily house dust mite sublingual immunotherapy tablet (HDM-SLIT tablet, 12 SQ-HDM dose).
- Placebo SLIT-tablet: Rhinitis/rhinoconjunctivitis rescue medication as needed, plus daily placebo sublingual immunotherapy tablet (Placebo SLIT-tablet).
Period: Overall Study
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Started (Randomised and treated) | 727 | 731
Completed (Completed IMP) | 688 | 705
Not Completed | 39 | 26
Not completed — Adverse Event | 18 | 6
Not completed — Lost to Follow-up | 2 | 3
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Reason stated as 'Other' in the case report form (CRF) | 7 | 7

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet | Total
Number analyzed (Participants) | 727 | 731 | 1458
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants had to be 5-11 years old at randomization
  years | 8.0 (1.9) | 8.0 (1.9) | 8.0 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 254 | 495
  Male | 486 | 477 | 963
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 19 | 45
  Not Hispanic or Latino | 688 | 697 | 1385
  Unknown or Not Reported | 13 | 15 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 3 | 4
  Race: Black or African American | 1 | 4 | 5
  Race: White | 722 | 714 | 1436
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Multiple | 1 | 3 | 4
  Race: Other | 1 | 7 | 8
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 20 | 38
  United States | 21 | 19 | 40
  Ukraine | 165 | 165 | 330
  Poland | 176 | 177 | 353
  Slovakia | 33 | 33 | 66
  Bulgaria | 91 | 90 | 181
  France | 2 | 1 | 3
  Lithuania | 47 | 47 | 94
  Germany | 8 | 9 | 17
  Russia | 163 | 166 | 329
  Spain | 3 | 4 | 7
Allergy history [Count of Participants; unit: Participants] — All participants had a medical history of HDM allergic rhinitis or rhinoconjunctivitis. However, since 1 participant in the 12 SQ-HDM group had 'rhinitis' entered in the wrong eCRF form, the data incorrectly suggests that 1 participant did not have rhinitis/rhinoconjunctivitis even though they did.
  Participants | 726 | 731 | 1457
Baseline sensitisations [Count of Participants; unit: Participants]
  House dust mite only | 337 | 360 | 697
  House dust mite and others | 390 | 371 | 761
Asthma status at baseline [Count of Participants; unit: Participants]
  Reported asthma | 267 | 290 | 557
  ICS use | 148 | 160 | 308

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Total Combined Rhinitis Symptom and Medication Score (TCRS) During the Primary Efficacy Assessment Period
Description: The primary endpoint in the trial was the average daily total combined rhinitis symptoms and medication score (TCRS) during the primary efficacy assessment period. The average daily TCRS evaluates the treatment effect based on the reduction in daily rhinitis symptoms and medication score (on a scale of 0-24). Higher scores indicate more severe symptoms and/or more use of rhinitis medication. The endpoint is calculated as the average score of all reported daily values during the 8-week primary efficacy assessment period. For example, if a subject reported 56 daily TCRS values, the primary endpoint is calculated as the average of those values.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants in the full analysis set with observations in the primary efficacy period.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 693 | 706
score on a scale | 3.4 (0.3) | 4.4 (0.3)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The average daily TCRS was analysed using a linear mixed effect (LME) model with square root transformation. The model includes the square root of the endpoint as response variable, treatment and cohort as fixed factors, the square root of the baseline value as a covariate, country/region within cohort as a random effect, and with different residual errors specified for each treatment. No missing data approach was applied; Test type: Superiority; p < 0.0001, Mixed Models Analysis — This endpoint was controlled for multiplicity using hierarchical testing; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.5 to 1.4] — Placebo vs. 12 SQ-HDM

2. Secondary Outcome: The Average Rhinitis Daily Symptom Score (DSS) During the Primary Efficacy Assessment Period
Description: The average rhinitis DSS evaluates the treatment effect based on the reduction in daily rhinitis symptom score (on a scale of 0-12). Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the 8-week primary efficacy assessment period. For example, if a subject reported 56 rhinitis DSS values, the endpoint is calculated as the average of those values.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants in the full analysis set with observations in the primary efficacy period
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 693 | 706
score on a scale | 1.5 (0.1) | 1.9 (0.1)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The average rhinitis DSS was analysed using a linear mixed effect (LME) model with square root transformation. The model includes the square root of the endpoint as response variable, treatment and cohort as fixed factors, the square root of the baseline value as a covariate, country/region within cohort as a random effect, and with different residual errors specified for each treatment. No missing data approach was applied; Test type: Superiority; p < 0.0001, Mixed Models Analysis — This endpoint was controlled for multiplicity using hierarchical testing; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.2 to 0.6] — Placebo vs. 12 SQ-HDM

3. Secondary Outcome: The Average Rhinitis Daily Medication Score (DMS) During the Primary Efficacy Assessment Period
Description: Average rhinitis DMS evaluates the treatment effect based on the reduction in daily rhinitis medication use (on a scale of 0-12). Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the 8-week primary efficacy assessment period. For example, if a subject reported 56 rhinitis DMS values, the endpoint is calculated as the average of those values.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants in the full analysis set with observations in the primary efficacy period.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 693 | 706
score on a scale | 1.4 (0.2) | 1.9 (0.2)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The average rhinitis DMS was analysed using a linear mixed effect (LME) model with square root transformation. The model includes the square root of the endpoint as response variable, treatment and cohort as fixed factors, the square root of the baseline value as a covariate, country/region within cohort as a random effect, and with different residual errors specified for each treatment. No missing data approach was applied; Test type: Superiority; p = 0.0016, Mixed Models Analysis — This endpoint was controlled for multiplicity using hierarchical testing; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.2 to 0.8]

4. Secondary Outcome: The Average Daily Total Combined Rhinoconjunctivitis Symptom and Medication Score (TCS) During the Primary Efficacy Assessment Period
Description: Average rhinoconjunctivitis TCS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis symptoms and medication use (on a scale of 0-38). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the 8-week primary efficacy assessment period. For example, if a subject reported 56 daily TCS values, the endpoint is calculated as the average of those values.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants in the full analysis set with observations in the primary efficacy period
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 693 | 706
score on a scale | 4.0 (0.4) | 5.2 (0.4)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; Test type: Superiority; p < 0.0001, Mixed Models Analysis — This endpoint was controlled for multiplicity using hierarchical testing; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [0.6 to 1.7] — Placebo vs.12 SQ-HDM

5. Secondary Outcome: The Average Rhinoconjunctivitis Daily Symptom Score (DSS) During the Primary Efficacy Assessment Period
Description: The average rhinoconjunctivitis DSS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis symptom score (on a scale of 0-18). Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the 8-week primary efficacy assessment period. For example, if a subject reported 56 rhinoconjunctivitis DSS values, the endpoint is calculated as the average of those values.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants in the full analysis set with observations in the primary efficacy period
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 693 | 706
score on a scale | 1.7 (0.1) | 2.2 (0.2)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The average rhinoconjunctivitis DSS was analysed using a linear mixed effect (LME) model with square root transformation. The model includes the square root of the endpoint as response variable, treatment and cohort as fixed factors, the square root of the baseline value as a covariate, country/region within cohort as a random effect, and with different residual errors specified for each treatment. No missing data approach was applied; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.3 to 0.7] — Placebo vs. 12 SQ-HDM

6. Secondary Outcome: The Average Rhinoconjunctivitis Daily Medication Score (DMS) During the Primary Efficacy Assessment Period
Description: Average rhinoconjunctivitis DMS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis medication use (on a scale of 0-20). Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the 8-week primary efficacy assessment period. For example, if a subject reported 56 rhinoconjunctivitis DMS values, the endpoint is calculated as the average of those values.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants in the full analysis set with observations in the primary efficacy period.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 693 | 706
score on a scale | 1.8 (0.2) | 2.4 (0.3)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The average rhinoconjunctivitis DMS was analysed using a linear mixed effect (LME) model with square root transformation. The model includes the square root of the endpoint as response variable, treatment and cohort as fixed factors, the square root of the baseline value as a covariate, country/region within cohort as a random effect, and with different residual errors specified for each treatment. No missing data approach was applied; Test type: Superiority; p = 0.0018, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.2 to 1.0] — Placebo vs. 12 SQ-HDM

7. Secondary Outcome: Overall Paediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) Score at the End of Trial
Description: The overall PRQLQ score measures the effect of rhinoconjunctivitis on participant's quality of life on a scale of 0-6. Higher scores indicate worse rhinoconjunctivitis-related quality of life.
Time Frame: Week leading up to visit 7 (at the end of the primary efficacy assessment period, after approximately 52-57 weeks of treatment)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 695 | 690
score on a scale | 0.8 (0.1) | 1.0 (0.1)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The overall PRQLQ score was analysed using a linear mixed effect (LME) model. The model includes the overall PRQLQ score as response variable, treatment and cohort as fixed factors, the baseline overall PRQLQ score as a covariate, country/region within cohort as a random effect, and with different residual errors specified for each treatment. No missing data approach was applied; Test type: Superiority; p < 0.0001, Mixed Models Analysis — This endpoint was controlled for multiplicity using hierarchical testing; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [0.1 to 0.2] — Placebo vs. 12 SQ-HDM

8. Secondary Outcome: The Average Asthma Daily Symptom Score (DSS) During the Primary Efficacy Assessment Period
Description: The average asthma DSS evaluates the treatment effect based on the reduction in daily asthma symptom score (on a scale of 0-12). Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the 8-week primary efficacy assessment period. For example, if a subject reported 56 asthma DSS values, the endpoint is calculated as the average of those values.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants with asthma in the full analysis set with observations in the primary efficacy period
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 251 | 280
score on a scale | 0.3 (0.0) | 0.4 (0.0)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The average asthma DSS was analysed using a linear mixed effect (LME) model with square root transformation. The model includes the square root of the endpoint as response variable, treatment and cohort as fixed factors, the square root of the baseline value as a covariate, country/region within cohort as a random effect, and with different residual errors specified for each treatment. No missing data approach was applied; Test type: Superiority; p = 0.0259, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [0.0 to 0.2] — Placebo vs. 12 SQ-HDM

9. Secondary Outcome: SABA Free Days During the Primary Efficacy Assessment Period
Description: The endpoint SABA free days evaluates the treatment effect based on the reduction in SABA use. The higher the proportion of SABA free days the higher the estimated probability of a participant having a day where they didn't use SABA.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants with asthma in the full analysis set with observations in the primary efficacy period
Measure: Number (95% Confidence Interval); unit: Probability (%) of a SABA free day
Groups:
- HDM SLIT-tablet (12 SQ-HDM): Rhinitis/rhinoconjunctivitis rescue medication as needed, plus daily house dust mite sublingual allergy immunotherapy tablet (HDM-SLIT tablet, 12 SQ-HDM dose).
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 251 | 280
Probability (%) of a SABA free day | 99.2 [98.6 to 99.6] | 98.6 [97.7 to 99.2]
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The odds of having a SABA free day was analysed using a generalised linear mixed model (GLMM) with a logit link function. The model included SABA free day (yes/no) as response variable, treatment and cohort as fixed effects, the baseline average asthma DSS as a covariate, the combined (country/region) variable within cohort and subject as random effects. Proportion is the estimated probability of having a day where a subject with asthma did not use SABA, odds ratio is (odds active/odds Placebo); Test type: Superiority; p = 0.0527, Generalised linear mixed model (GLMM); Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.0 to 3.3] — Odds ratio is (odds 12 SQ-HDM / odds Placebo)

10. Secondary Outcome: Weekly Number of Puffs of As-needed SABA Use During the Primary Efficacy Assessment Period
Description: Average weekly number of puffs of as-needed SABA use evaluates the treatment effect based on the reduction in the use of asthma reliever medication (SABA), and is calculated as 7 times the average of the daily number of puffs of as-needed SABA use. Higher values indicate more medication use.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants with asthma in the full analysis set with observations in the primary efficacy period.
Measure: Mean (Standard Error); unit: weekly number of puffs
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 251 | 280
weekly number of puffs | 1.0 (0.2) | 1.5 (0.2)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The endpoint was analysed using a linear mixed effect (LME) model. The model includes the endpoint as response variable, treatment and cohort as fixed factors, the baseline value as a covariate, country/region within cohort as a random effect, and with different residual errors specified for each treatment. No missing data approach was applied; Test type: Superiority; p = 0.1256, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.1 to 1.0] — Placebo vs. 12 SQ-HDM

11. Secondary Outcome: Rhinitis Mild Days During the Primary Efficacy Assessment Period
Description: The endpoint rhinitis mild days evaluates the treatment effect based on days when participants have no symptoms or mild symptoms and no medication use. The higher the proportion of rhinitis mild days the higher the estimated probability of a participant having a rhinitis mild day.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants with asthma in the full analysis set with observations in the primary efficacy period
Measure: Number (95% Confidence Interval); unit: Probability (%) of a rhinitis mild day
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 693 | 706
Probability (%) of a rhinitis mild day | 31.8 [22.6 to 42.8] | 20.9 [14.2 to 29.7]
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The odds of having a rhinitis mild day was analysed using a generalised linear mixed model (GLMM) with a logit link function. The model included the endpoint (yes/no) as response variable, treatment and cohort as fixed effects, the baseline average rhinitis TCRS as a covariate, the combined (country/region) variable within cohort and subject as random effects. Proportion is the estimated probability of having a day with no or mild rhinitis symptoms, odds ratio is (odds 12 SQ-HDM / odds Placebo); Test type: Superiority; p = 0.0008, Generalised linear mixed model (GLMM); Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.3 to 2.5] — Odds ratio is (odds 12 SQ-HDM / odds Placebo)

12. Secondary Outcome: Rhinitis Exacerbation Days During the Primary Efficacy Assessment Period
Description: The endpoint rhinitis exacerbation days evaluates the treatment effect based on days when participants have severe symptoms. The higher the proportion of rhinitis mild days the higher the estimated probability of a participant having a rhinitis exacerbation day.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants in the full analysis set with observations in the primary efficacy period
Measure: Number (95% Confidence Interval); unit: Probability (%) of a rhinitis exace. day
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 693 | 706
Probability (%) of a rhinitis exace. day | 2.5 [1.7 to 3.6] | 4.4 [3.1 to 6.2]
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM); The odds of having a rhinitis exacerbation day was analysed using a generalised linear mixed model (GLMM) with a logit link function. The model included the endpoint (yes/no) as response variable, treatment and cohort as fixed effects, the baseline average rhinitis DSS as a covariate, the combined (country/region) variable within cohort and subject as random effects. Proportion is the estimated probability of having a rhinitis exacerbation day, odds ratio is (odds 12 SQ-HDM / odds Placebo); Test type: Superiority; p < 0.0001, Generalised linear mixed model (GLMM); Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.4 to 0.7] — Odds ratio is (odds 12 SQ-HDM / odds Placebo)

13. Secondary Outcome: Average Rhinitis Combined Symptom and Medication Score (CSMS) During the Primary Efficacy Assessment Period
Description: Average rhinitis CSMS evaluates the treatment effect based on the reduction in daily rhinitis symptoms and/or medication use. For this endpoint, the rhinitis symptoms and medication use were scored using an alternative method as recommended by EAACI (European Academy of Allergy & Clinical Immunology) (on a scale of 0-5). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the 8-week primary efficacy assessment period. For example, if a subject reported 56 rhinitis CSMS values, the endpoint is calculated as the average of those values.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants in the full analysis set with observations in the primary efficacy period.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 693 | 706
score on a scale | 0.8 (0.1) | 1.0 (0.1)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The average rhinitis CSMS was analysed using a linear mixed effect (LME) model with square root transformation. The model includes the square root of the endpoint as response variable, treatment and cohort as fixed factors, the square root of the baseline value as a covariate, country/region within cohort as a random effect, and with different residual errors specified for each treatment. No missing data approach was applied; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [0.1 to 0.3] — Placebo vs. 12 SQ-HDM

14. Secondary Outcome: Average Rhinoconjunctivitis Combined Symptom and Medication Score (CSMS) During the Primary Efficacy Assessment Period
Description: Average rhinoconjunctivitis CSMS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis symptoms and/or medication use. For this endpoint, the rhinoconjunctivitis symptoms and medication use were scored using an alternative method as recommended by EAACI (European Academy of Allergy & Clinical Immunology) (on a scale of 0-5). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the 8-week primary efficacy assessment period. For example, if a subject reported 56 rhinoconjunctivitis CSMS values, the endpoint is calculated as the average of those values.
Time Frame: 8 weeks (primary efficacy assessment period), which started 44-49 weeks after initiation of IMP
Population: Participants in the full analysis set with observations in the primary efficacy period.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 693 | 706
score on a scale | 0.7 (0.1) | 0.9 (0.1)
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The average rhinoconjunctivitis CSMS was analysed using a linear mixed effect (LME) model with square root transformation. The model includes the square root of the endpoint as response variable, treatment and cohort as fixed factors, the square root of the baseline value as a covariate, country/region within cohort as a random effect, and with different residual errors specified for each treatment. No missing data approach was applied; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [0.1 to 0.3] — Placebo vs. 12 SQ-HDM

15. Secondary Outcome: House Dust Mite Specific IgE
Description: House dust mite specific IgE reflects the allergen-specific allergy immunotherapy-induced immune modulation
Time Frame: Change from screening to the end of trial (after approximately 52-57 weeks of treatment)
Population: Participants from Canada and Poland in the full analysis set with observations
Measure: Mean (Standard Deviation); unit: log10 transformed kU/L
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 178 | 184
log10 transformed kU/L
  Dermatophagoides pteronyssinus specific IgE | 0.2 (0.3) | 0.0 (0.2)
  Dermatophagoides farinae specific IgE | 0.3 (0.3) | 0.0 (0.2)

16. Secondary Outcome: House Dust Mite Specific IgG4
Description: House dust mite specific IgG4 reflects the allergen-specific allergy immunotherapy-induced immune modulation
Time Frame: Change from screening to the end of trial (after approximately 52-57 weeks of treatment)
Population: Participants from Canada and Poland in the full analysis set with observations
Measure: Mean (Standard Deviation); unit: log10 transformed mg/L
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 178 | 184
log10 transformed mg/L
  Dermatophagoides pteronyssinus specific IgG4 | 0.6 (0.4) | 0.0 (0.1)
  Dermatophagoides farinae specific IgG4 | 0.7 (0.4) | 0.0 (0.2)

17. Secondary Outcome: Total IgE
Description: The change in total IgE was measured from screening to the end of trial.
Time Frame: Change from screening to the end of trial (after approximately 52-57 weeks of treatment)
Population: Participants from Canada and Poland in the full analysis set with observations
Measure: Mean (Standard Deviation); unit: log10 transformed kU/L
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 178 | 183
log10 transformed kU/L | 0.2 (0.3) | 0.0 (0.2)

18. Secondary Outcome: House Dust Mite IgE-Blocking Factor
Description: The IgE-blocking factor assesses the effect of serum components (including IgE-blocing antibodies known to be induced by allergy immunotherapy) competing with IgE for binding to allergen. IgE-blocking factor is calculated as 1-(S/T), where S is the amount of allergen-specific IgE bound to allergen in the (possible) presence of competing components, and where T is the total amount of allergen-specific IgE capable of binding to allergen when all competing antibodies/components have been washed off. IgE-blocking factor values closer to 0 indicate the presence of fewer IgE-blocking components and values closer to 1 indicate that more IgE is blocked from binding to the allergen.
Time Frame: Change from screening to the end of trial (after approximately 52-57 weeks of treatment)
Population: Participants from Canada and Poland in the full analysis set with observations
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 103 | 140
unitless | 0.4 (0.3) | -0.0 (0.1)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from consent until the last follow-up phone contact with the participant (from V1 to TC3 (telephone call 3), for approximately 54-59 weeks).
Description: Treatment emergent AEs (TEAEs) are displayed (these were AEs starting on/after time of first IMP and no later than 7 days after last day of IMP). For the first 28 days of treatment, the presence/absence of 15 specific symptoms, identified as local side effects of sublingual immunotherapy (solicited events), were captured in an eDiary. Solicited events were evaluated by the investigator and reported in the eCRF as AEs as per their discretion. TEAEs from the eCRF are presented.
Groups:
- HDM SLIT-tablet (12 SQ-HDM): Rhinitis/rhinoconjunctivitis rescue medication and asthma controller/reliever medication as needed, plus daily house dust mite sublingual allergy immunotherapy tablet (HDM-SLIT tablet, 12 SQ-HDM dose).
- Placebo SLIT-tablet: Rhinitis/rhinoconjunctivitis rescue medication and asthma controller/reliever medication as needed, plus daily placebo sublingual allergy immunotherapy tablet (Placebo SLIT-tablet).
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
All-Cause Mortality (participants affected / at risk) | 0/727 | 0/731
Serious Adverse Events (participants affected / at risk) | 16/727 | 6/731
Other Adverse Events (participants affected / at risk) | 608/727 | 534/731
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDM SLIT-tablet (12 SQ-HDM) (N=727) | Placebo SLIT-tablet (N=731)
Gastroenteritis norovirus (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pseudomonas bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDM SLIT-tablet (12 SQ-HDM) (N=727) | Placebo SLIT-tablet (N=731)
Oral pruritus (Gastrointestinal disorders) | 419 (1149) | 185 (425)
Abdominal pain upper (Gastrointestinal disorders) | 243 (512) | 164 (320)
Lip swelling (Gastrointestinal disorders) | 151 (282) | 38 (63)
Glossodynia (Gastrointestinal disorders) | 142 (313) | 41 (54)
Nausea (Gastrointestinal disorders) | 135 (260) | 81 (125)
Mouth swelling (Gastrointestinal disorders) | 99 (210) | 27 (41)
Swollen tongue (Gastrointestinal disorders) | 99 (203) | 20 (29)
Diarrhoea (Gastrointestinal disorders) | 95 (151) | 74 (107)
Mouth ulceration (Gastrointestinal disorders) | 93 (162) | 53 (80)
Tongue ulceration (Gastrointestinal disorders) | 50 (82) | 27 (34)
Vomiting (Gastrointestinal disorders) | 48 (76) | 33 (38)
Tooth loss (Gastrointestinal disorders) | 40 (66) | 35 (61)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 401 (1072) | 236 (504)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 68 (134) | 22 (33)
Asthma (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 38 (49)
Nasopharyngitis (Infections and infestations) | 185 (250) | 164 (206)
COVID-19 (Infections and infestations) | 38 (38) | 38 (38)
Pharyngitis (Infections and infestations) | 38 (44) | 37 (49)
Bronchitis (Infections and infestations) | 36 (42) | 45 (52)
Upper respiratory tract infection (Infections and infestations) | 22 (29) | 37 (53)
Ear pruritus (Ear and labyrinth disorders) | 242 (547) | 135 (299)
Taste disorder (Nervous system disorders) | 123 (213) | 116 (218)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication can be made before the primary publication. PI shall provide Sponsor (S) with a copy of any publication or presentation 60 days before submission/public disclosure. S can require changes or non-publication of the article, if appropriate. Upon S request, the PI must delay the publication, presentation or public disclosure for an additional 120 days to permit S to apply for a patent application. Any other public statements regarding the trial requires prior written consent from S.

DOCUMENTS (2):
  • Study Protocol (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT04145219/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT04145219/SAP_001.pdf